CLINICAL TRIAL: NCT00619242
Title: A Pilot Study of the Effect of Sorafenib on Molecular Biomarkers in Barrett's Esophagus With High Grade Dysplasia
Brief Title: The Effects of Sorafenib on Molecular Barrett's Esophagus Cancer
Acronym: Barrett's
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Chicago (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14374B
Record Dates: First submitted 2008-02-06; First posted 2008-02-20 (Estimated); Results first posted 2013-10-21 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-02

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sorafenib (Experimental): sorafenib 2 tablets by mouth
  Interventions: Drug: sorafenib

INTERVENTIONS:
Drug: sorafenib — 2 tablets with water by mouth twice a day for two weeks.

SUMMARY:
To determine whether sorafenib is able to change pre-cancerous cells in a way that we believe is important in the progression of cancer.

DETAILED DESCRIPTION:
To characterize the effects of sorafenib on specific molecular markers in patients with Barrett's esophagus and high grade intraepithelial neoplasia (HGIN) or carcinoma in situ (CIS).

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0-2
* Life expectancy of greater than 12 months
* No prior history of esophageal surgery or endoscopic treatment of dysplasia
* No prior exposure to sorafenib
* Patients may not be receiving any other investigational agents or any concomitant antineoplastic therapy, with the exception of androgen ablating agents (for patients with prior prostate cancer)
* Age 18 years.
* Patients must have adequate organ and marrow function as defined below:

  * hemoglobin: 8.5 g/dL
  * absolute neutrophil count: 1,500/L
  * platelets: 100,000/L (greater than 35,000/L without transfusion for less than 1 X the institutional upper limit of normal)
  * creatinine less than 1.5 X institutional upper limit of normal
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* A patient will be withdrawn from the study if any of the following events occur while on therapy:

  * Interruption of scheduled therapy for greater than 7 days
  * Intolerable adverse effects which are judged by the investigator to be either physically or psychologically detrimental to the patient
  * Patient decision to discontinue treatment
  * Pregnancy
  * Patient non-compliance with therapy administration
  * Grade 3 or 4 NCI-CTC toxicity attributable to sorafenib
  * Treatment with other chemotherapeutic or investigational anti-neoplastic drugs
  * Disease progression
* HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with sorafenib.Appropriate studies will be undertaken in patients receiving combination anti-retroviral therapy when indicated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated and opened to accrual 06/19/2006. the study was terminated 7/17/2009. Subjects were seen in the University of Chicago outpatient clinics.
Pre-assignment Details: Subjects must have histologically confirmed Barrett's esophagus with high-grade intraepithelial neoplasia (HGIN) or carcinoma in situ (CIS) on prior endoscopy within the previous 12 months.
Groups:
- Sorafenib: Sorafenib 400mg BID
Period: Overall Study
Arm/Group | Sorafenib
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Ki-67
Description: Biomarker. Change in Ki-67 staining between pre- and on-therapy biopsies in patients with Barrett's esophagus.
Time Frame: Two weeks
Population: The 3 subjects underwent therapy without complications however the study was terminated due to low accrual.
Arm/Group | Sorafenib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sorafenib
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes